CLINICAL TRIAL: NCT01986296
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound Treatment of Medication-Refractory OCD
Brief Title: ExAblate Treatment of Medication Refractory Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCD001
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Medication-refractory Obsessive Compulsive Disorder (OCD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExAblate Treatment (Experimental)
  Interventions: Device: ExAblate Transcranial MRgFUS System

INTERVENTIONS:
Device: ExAblate Transcranial MRgFUS System — Treatment with the ExAblate Transcranial MRgFUS System.

SUMMARY:
The goal of this prospective, non-randomized, single-arm, single site, feasibility study is to develop and collect data to evaluate the safety and initial effectiveness of this treatment using this ExAblate transcranial System in the treatment of Medication-Refractory OCD.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and initial effectiveness of MRI-guided focused ultrasound thermal ablation of a designated area in the brain of patients suffering from medication-refractory OCD, using the ExAblate transcranial system.

The ExAblate system is a medical device that involves a focused ultrasound system and an MRI scanner. ExAblate delivers a pulse of focused ultrasound energy, or sonication, to the targeted tissue. For OCD Patients: one or more thermal lesion will be created on one of the following targets: Anterior cingulate cortex, Anterior Limb of internal Capsule, Ventral Striatum or Subgenual Cingulate Cortex.

The treatment begins with a series of standard diagnostic MR images to identify the location and shape of tumor to be treated. The ExAblate computer uses the physician's designation of the target volume to plan the best way to cover the target volume with small spots called "sonications". These treatment spots are cylinder shaped. Their size depends on sonication power and duration. During the treatment, a specific MR scan, which can be processed to identify changes in tissue temperature, provides a thermal map of the treatment volume to confirm the therapeutic effect. The thermal map is used to monitor the treatment in progress, and confirm that the ablation is proceeding according to plan, thus closing the therapy loop.

The ExAblate transcranial operates a helmet-shaped transducer (currently utilizing 1000-element phased array transducer) positioned above the subject head. The ExAblate transcranial system also includes means to immobilize the subject head, cool the interface water, and software for CT analysis and phase correction computation.

After informed consent and screening, eligible subjects will proceed to the treatment. All subjects will be followed at Day 1, 7 days, 1 month, 6 months and 1, 2 and 3 years. At follow up visits, patients will be evaluated for general health, neurological changes (including MMSE exam),and efficacy measurements as well as for device/procedure related adverse events that may have occurred during the follow-up period. Six (6) month and 1, 2 and 3 year follow up visits will also include Full Battery Cognitive/Neurological Testing.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, between 18 and 65 years, inclusive
2. Subjects who are able and willing to give consent and able to attend all study visits
3. OCD refractory to adequate trials of medication and behavioral therapy by psychiatrist (more than 12 weeks at the maximum tolerated dose with more than two types of serotonin reuptake inhibitors).
4. Designated Ablation Targets can be target by the ExAblate device. Designated Ablation Targets must be apparent on MRI such that targeting can be performed with direct visualization.
5. Able to communicate sensations during the ExAblate MRgFUS treatment
6. Definitive diagnosis of OCD, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorder fourth edition (DSM-IV), with disease duration of more than 3 years, with diagnosed psychosocial dysfunction. (The diagnosis of OCD would be done by psychiatrist)
7. A score on the Y-BOCS of more than 28.
8. OCD medication regimen is stable for at least 30 days before enrolment
9. Patients with diagnosed psychosocial dysfunction influenced by OCD

Exclusion Criteria:

1. Patients with unstable cardiac status including:

   1. Unstable angina pectoris on medication
   2. Patients with documented myocardial infarction within last 40 days to protocol entry
   3. Congestive heart failure NYHA Class IV
2. Patients exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period:

   * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
   * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
   * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
   * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
3. Severe hypertension (diastolic BP > 100 on medication)
4. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
5. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium/Magnevist) including advanced kidney disease
6. Patients receiving dialysis
7. History of abnormal bleeding and/or coagulopathy
8. Receiving anticoagulant (e.g. Warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of scheduled focused ultrasound procedure
9. Active or suspected, acute or chronic uncontrolled infection or known life-threatening systemic disease
10. History of intracranial hemorrhage
11. Cerebrovascular disease (multiple CVA or CVA within 6 months)
12. Evidence for calcifications that might interfere with treatment safety (per CT)
13. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
14. Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
15. Patients unable to communicate with the investigator and staff
16. Presence of any other neurodegenerative disease like Parkinson-plus syndromes suspected on neurological examination. These include:

    1. Multisystem atrophy
    2. Progressive supranuclear palsy
    3. Dementia with Lewy bodies
    4. Alzheimer's disease
17. Subjects diagnosed with idiopathic Parkinson's disease.
18. Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
19. History of immunocompromise, including patient who are HIV positive
20. Patients with a history of seizures within the past year
21. Patients with risk factors for intraoperative or postoperative bleeding:

    1. Platelet count less than 100,000 per cubic millimeter
    2. PT > 14
    3. PTT > 36
    4. INR > 1.3
    5. Documented coagulopathy
    6. Patients receiving medications that are known to induce or contribute to Hemorrhages
22. Patients with any types of brain tumors, including metastases
23. Any illness that in the investigator's opinion preclude participation in this study
24. Pregnancy or lactation
25. Patients who have had deep brain stimulation or a prior stereotactic ablation of Designated Ablation Target
26. OCD medication regimen is not stable for at least 30 days before enrolment
27. Legal incapacity or limited legal capacity
28. Subjects with remarkable atrophy and poor healing capacity of the scalp (> 30% of the skull area traversed by the sonication pathway)
29. Are participating or have participated in another clinical trial in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the ExAblate Transcranial MRgFUS treatment of medication-refractory OCD | Participants will be followed from the date of treatment until study completion, up to 36 months
  Effectiveness of the ExAblate Transcranial MR-guided Focused Ultrasound (MRgFUS) treatment of medication-refractory OCD will be determined using the Yale-Brown Obsessive-Compulsive Disorder Scale (Y-BOCS), Hamilton Depression Rating Scale (HAM-D), and Hamilton Anxiety Rating Scale (HAM-A) from examinations at baseline and through 6-Months post-ExAblate treatment.

SECONDARY OUTCOMES:
Device or procedure related Adverse Events reported | 36 month
  Safety of the ExAblate transcranial treatment will be determined by an evaluation of the incidence and severity of device and procedure related complications from the first / treatment day visit through the 6-Months post-treatment time point. All Adverse Events (AEs) will be reported and categorized by investigators as definitely, probably, possibly, or unrelated to the device, procedure, or post-surgical changes in neurological status. Alternative treatments resulting from post-surgical changes in neurological status will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Chang, Prof., Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Medical Center, Seoul, South Korea

REFERENCES:
- See also: Sponsor website — http://www.insightec.com